CLINICAL TRIAL: NCT03894007
Title: Improving Pre-operative Systemic Therapy for Human Epidermal Growth Factor Receptor 2 (HER2) Amplified Breast Cancer Part of a Platform of Translational Phase II Trials Based on Molecular Subtypes
Brief Title: Improving Pre-operative Systemic Therapy for Human Epidermal Growth Factor Receptor 2 (HER2) Amplified Breast Cancer
Acronym: PREDIXIIHER2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Security and effect data from another ongoing study.
Sponsor: Renske Altena (Other)
Responsible Party: Sponsor-Investigator, Renske Altena, MD, PhD. Principal Investigator., Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIX II HER2; 2018-004457-24 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-28 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Early-stage Breast Cancer; HER2-positive Breast Cancer
Keywords: Neoadjuvant therapy; PD-L1 positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Epirubicin; Cyclophosphamide; atezolizumab; Ado-Trastuzumab Emtansine; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Both arms start with four cycles of docetaxel/paklitaxel+carboplatin+trastuzumab+pertuzumab. Thereafter arm A receives three cycles of epirubicin+cyclophosphamide+atezolizumab and arm B receives epirubicin+cyclophosphamide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A: Experimental (Experimental): Four courses of docetaxel or paclitaxel + carboplatin + trastuzumab sc + pertuzumab given every third week followed by three courses of epirubicin + cyclophosphamide + atezolizumab. In total seven courses of preoperative treatment. Response evaluations after course four.
  Postoperatively, if pathologic complete response, patients receive 14 courses of adjuvant trastuzumab every third week. If no pCR patients receive 14 courses of T-DM1 every third week.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Atezolizumab; Drug: Trastuzumab emtansine; Drug: Paclitaxel
- B: Standard (Active Comparator): Four courses of docetaxel or paclitaxel + carboplatin + trastuzumab sc + pertuzumab given every third week followed by three courses of epirubicin + cyclophosphamide. In total seven courses of preoperative treatment. Response evaluations after course four.
  Postoperatively, if pathologic complete response patients receive 14 courses of adjuvant trastuzumab (combined with pertuzumab in case of high-risk disease features) every third week. If no pCR patients receive 14 courses of T-DM1 every third week.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Trastuzumab emtansine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 iv, escalated to 100 mg/m2 if tolerated, day 1 every third week, 4 courses preoperatively.
Drug: Carboplatin — AUC 6 iv, day 1 every third week, 4 courses preoperatively.
Drug: Trastuzumab — 600 mg sc, day 1 every third week, 4 courses preoperatively. 14 courses postoperatively if complete response.
  Other Names: Herceptin
Drug: Pertuzumab — 840 mg iv starting dose, thereafter 420 mg, day 1 every third week. 14 courses postoperatively if complete response in patients with baseline high risk tumours.
  Other Names: Perjeta
Drug: Epirubicin — 90 mg/m2 iv, escalated to 100 mg/m2 if tolerated, day 1 every third week, 3 courses preoperatively
Drug: Cyclophosphamide — 600 mg/m2 iv, day 1 every third week, 3 courses preoperatively
Drug: Atezolizumab — 840 mg iv, day 1 every third week, 3 courses preoperatively if randomised to arm A.
  Other Names: Tecentriq
  Arms: A: Experimental
Drug: Trastuzumab emtansine — 3.6 mg/kg iv, day 1 every third week, 14 courses postoperatively if not complete response.
  Other Names: Kadcyla
Drug: Paclitaxel — 80 mg/m2 iv, day 1 weekly, 12 weeks (4 cycles), in case of (anticipated) unmanageable toxicity related to docetaxel.

SUMMARY:
This is a phase 2 study evaluating medical treatment before surgery in HER2-amplified early breast cancer patients. Patients receive chemotherapy with HER2-targeted antibodies and are randomised to receive the checkpoint inhibitor atezolizumab or not.

DETAILED DESCRIPTION:
The primary aim is to investigate whether the rate of pCR, after optimal neoadjuvant anti-HER2 based systemic therapy, can be increased by addition of atezolizumab.

Secondary aims are to assess safety and tolerability of this treatment combination, and to identify therapy predictive factors for the anti-HER2 monoclonal antibodies trastuzumab and pertuzumab plus-minus atezolizumab with a backbone of chemotherapy, using modern molecular biological investigational procedures with analyses by repeated biopsies from an intra-patient longitudinal study design.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PD-L1 expression ≥1% on tumour cells and/or TILs (prescreening phase)
* Able to provide written informed consent
* Female gender
* Patients with breast cancer confirmed by histology, characterised by immunohistochemistry for ER, PR, HER2 and proliferation marker.
* HER2 amplification, IHC 3+ and preferably confirmed by ISH
* Tumor and blood samples available.
* Age 18 years or older. Elderly patients in adequate condition for the planned therapy, which may be supported by a geriatric assessment (according to ASCO guideline; Mohile et al, JCO 2018)
* Primary breast cancer >20 mm in diameter or verified lymph node metastases
* Adequate bone marrow, renal and hepatic functions (see Table 1)
* LVEF ≥50%
* ECOG performance status 0-1

Exclusion Criteria:

* Distant metastases without chance to cure, including node metastases in the contralateral thoracic region or in the mediastinum. An exception is presence of at most 2 morphologically characterized well-defined distant metastases accessible for stereotactic radiotherapy, provided that this treatment is available at the participating centre.
* Other malignancy diagnosed within the last five years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix
* Patients in child-bearing age without adequate contraception
* Pregnancy or lactation
* Uncontrolled hypertension, heart-, liver-, or kidney-diseases or other medical/psychiatric disorders.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study. Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) are permitted provided that they meet the following conditions:

    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids
    * No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids).
* Vaccination with a live vaccine within 30 days of the first dose of study treatment
* A known history of Human Immunodeficiency Virus (HIV) infection, hepatitis B (HBsAg reactive) or hepatitis C (HCV RNA detected) infection or active tuberculosis.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study
  * Patients with a history of allergic reaction to IV contrast requiring steroid pre- treatment should have baseline and subsequent tumor assessments performed using MRI.
  * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
* Hypersensitivity to atezolizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of pathological objective response to primary medical treatment | At surgery 2-3 weeks after the last (of 7) cycles of neo-adjuvant systemic therapy.
  Efficacy measure at surgery that is performed 2-3 weeks after 7 cycles (each cycle lasts 21 days) of preoperative treatment.

SECONDARY OUTCOMES:
Objective response rate | After the 4th and 7th cycle (each cycle is 21 days)
  Proportion of patients with reduction in tumour burden ≥30% according to RECIST
Distant disease-free survival | During the study period up to 10 years
  Time from randomisation to distant metastases or death due to breast cancer
Event-free survival | During the study period up to 10 years
  Time from randomisation to breast cancer relapse, contralateral breast cancer, other malignant neoplasms, or death from any cause
Overall survival | During the study period up to 10 years
  Time from randomisation to death from any cause
Rate of breast conserving surgery | At surgery
  Rate
Incidence of treatment-emergent adverse events (Safety) | During the 18-week period of treatment and until 30 days after termination and during the follow-up period up to ten years
  Rate of grade 3-4 toxicity, rate of % of discontinuation of study medication due to toxicity, rate of AE's of special interest
Differences in PROMs according to EORTC C30 | At baseline, after cycle 4 (a cycle is 21 days), after cycle 7 (a cycle is 21 days), 2 months, 1 year and 5 years after surgery
  Health related Quality of Life using the EORTC C30 scale (EORTC Quality of Life questionnaire C30)
Differences in PROMs according to EORTC BR23 | At baseline, after cycle 4 (a cycle is 21 days), after cycle 7 (a cycle is 21 days), 2 months, 1 year and 5 years after surgery
  Health related Quality of Life using the EORTC BR23 scale (EORTC Quality of Life breast specific questionnaire BR23)
Differences in objective cognitive function | At baseline, 3 months after surgery, one and five year after treatment start
  Assessed by an online neuropsychological test (Amsterdam Cognition Scan, validated for use in breast cancer patients [Feenstra et al, J Clin Exp Neuropsychol. 2018 Apr;40(3):253-273. ])
Treatment prediction, PD-L1 | At baseline, after the 4th cycle (each cycle is 21 days), at surgery and annually during the post-surgical follow-up period up to five years
  % of Programmed Death Ligand 1 expressing cells [tumour cells and tumour infiltrating lymphocytes]
Treatment prediction, TMB | At baseline, after the 4th cycle (each cycle is 21 days), at surgery and annually during the post-surgical follow-up period up to five years
  Tumour-mutational burden (total number of nonsynonymous mutations per coding area of a tumor genome)
Treatment prediction, TILs | At baseline, after the 4th cycle (each cycle is 21 days), at surgery and annually during the post-surgical follow-up period up to five years
  Percentage of tumour infiltrating lymphocytes
Treatment prediction, composition of faeces microbiome | At baseline, after 7th cycle (each cycle is 21 days) before surgery, and one year after surgery
  Composition of bacterial strains in gastro-intestinal flora (% of different strains measured with DNA/RNA analysis and in microbiotic culture)
Differences in PROMs | At baseline, after cycle 4 (each cycle is 21 days), after cycle 7 (each cycle is 21 days), 2 months, 1 year and 5 years after surgery
  Symptoms using the Memorial Symptoms Assessment Scale (MSAS). The 32-item MSAS scale includes occurrence, frequency, severity, and distress associated with each symptom using four- and five-point rating scales. Symptom burden is calculated as the average of frequency, severity and distress of each symptom. Higher scores indicates higher symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Renske Altena, MD, PhD, Principal Investigator — Karolinska University Hospital; Jonas Bergh, MD, PhD, Study Director — Karolinska Institutet
Locations (8):
- Sweden (8):
  - Sahlgrenska universitetssjukhuset, Gothenburg
  - Skånes universitetssjukhus, Malmo
  - Örebro universitetssjukhus, Örebro
  - Karolinska universitetssjukhuset, Stockholm
  - S:t Görans sjukhus, Stockholm
  - Södersjukhuset, Stockholm
  - Länssjukhuset Sundsvall, Sundsvall
  - Norrlands universitetssjukhus, Umeå